CLINICAL TRIAL: NCT00571415
Title: Image-guided Adaptive Radiotherapy for Cervix Cancer: Patient Image Acquisition
Status: Terminated | Type: Observational
Why Stopped: Due to competing studies no further subjects could be recruited.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM10390; P01CA116602 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Cervix Cancer
Keywords: Image guided adaptive radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cervix cancer patients

SUMMARY:
Within this study patient data are collected from different imaging and motion monitoring devices that will be used to develop and test strategies for image-guided adaptive radiotherapy in cervix cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of cervix cancer
* Prescription of radiation treatment to the primary cancer

Exclusion Criteria:

* Prior radiation treatment to the pelvis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospital clinic
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Increase in therapeutic ratio | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Williamson, PhD, Principal Investigator — Virginia Commonwealth University, Department of Radiation Oncology; Jeffrey F Williamson, PhD, Study Director — VCU, Richmond, VA
Locations (1):
- Viriginia Commonwealth University, Department of Radiation Oncology, Richmond, Virginia, United States